CLINICAL TRIAL: NCT03991858
Title: Implementation of Telerehabilitation as an Innovative Modality of Patient Follow-up on the Waiting List of the External Rehabilitation Clinic of the CIUSSS de l'Estrie-CHUS.
Brief Title: Implementation of Telerehabilitation as Modality of Patient Follow-up on the Waiting List of a Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Ministère de l'Économie, de la Science et de l'Innovation (Unknown)
Responsible Party: Principal Investigator, Michel Tousignant, Principal investigator, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-2919
Record Dates: First submitted 2019-05-02; First posted 2019-06-19 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Rehabilitation; Orthopedic Disorder
Keywords: Rehabilitation; Telerehabilitation; Waiting list; follow-up
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone follow-up (Other): Phone follow-up initiated by the health care professional one month after the initial evaluation at the external rehabilitation clinic.
  Interventions: Other: Phone call follow-up
- Telerehabilitation follow-up (Experimental): Telerehabilitation follow-up initiated by the health care professional one month after the initial evaluation at the external rehabilitation clinic.
  Interventions: Other: Telerehabilitation follow-up

INTERVENTIONS:
Other: Phone call follow-up — A physical therapist made a phone call to the patient one month after his/her initial evaluation at the external rehabilitation clinic
  Arms: Phone follow-up
Other: Telerehabilitation follow-up — A physical therapist made a direct follow-up through telerehabilitation to the patient one month after his/her initial evaluation at the external rehabilitation clinic
  Arms: Telerehabilitation follow-up

SUMMARY:
This study responds to the need to validate the feasibility and effectiveness of a telerehabilitation home monitoring program for users receiving a preliminary assessment while waiting for rehabilitation services at the outpatient physiotherapy clinic. The specific objectives are as followed: 1) Evaluate the implementation of telerehabilitation monitoring (TELE-FOLLOW-UP); 2) Evaluate the effectiveness of TELE-FOLLOW-UP compared to the usual phone call; 3) Evaluate user satisfaction for these two modes of service delivery; 4) Identify facilitators and barriers to the implementation of TELE-FOLLOW-UP. In order to meet the objectives of the study, mixed methods will be used. A randomized clinical trial will be used to achieve objectives 1, 2 and 3. The investigators plan to recruit 142 patients. Two groups will be formed: 1) TELE-FOLLOW-UP group: users who will receive follow-up by telerehabilitation; 2) PHONE-FOLLOW-UP group: those who will receive follow-up by a phone call.

DETAILED DESCRIPTION:
Rational : The rehabilitation service offered at the Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke (CIUSSS de l'Estrie - CHUS) for non-hospitalized patients is performed in outpatient clinics. However, the demand for this service far exceeds the supply, so the take-up time is very long. Recognizing the threatened short-term accessibility, this outpatient clinic has put in place an initial assessment for any service request. The goal is to conduct a preliminary assessment of the condition of the user to teach an exercise and education program. In addition, sporadic monitoring is recommended to promote the effectiveness of the intervention.

To date, the follow-up of this preliminary assessment is done by a phone call from the professional to the patient one month later. However, it is noted that this type of monitoring is not optimal for various reasons, in particular because of the absence of visual contact with the user to allow appropriate feedback from the professional on the exercise execution. In this context, the possibility of having a follow-up by a physiotherapist using telerehabilitation, an application of information technologies allowing a synchronous auditory and visual link, would be an innovative way of increasing the effectiveness of the intervention. This study therefore responds to the need to validate the feasibility and effectiveness of a telerehabilitation home monitoring program for users receiving a preliminary assessment while waiting for physiotherapist at the outpatient physiotherapy clinic. The results of this study will be relevant to clinicians and managers and will undeniably influence the provision of rehabilitation services.

Objectives: The specific objectives are as followed: 1) Evaluate the implementation of telerehabilitation monitoring (TELE-FOLLOW-UP); 2) Evaluate the effectiveness of TELE-FOLLOW-UP compared to the usual phone call; 3) Evaluate user satisfaction for these two modes of service delivery; 4) Identify facilitators and barriers to the implementation of TELE-FOLLOW-UP.

Methodology : In order to meet the objectives of the study, mixed methods will be used. A randomized clinical trial will be used to achieve objectives 1, 2 and 3. The investigators plan to recruit 142 patients. Two groups will be formed: 1) TELE-FOLLOW-UP group: users who will receive follow-up by telerehabilitation; 2) PHONE-FOLLOW-UP group: those who will receive follow-up by a phone call. In order to complete Objective 4, a qualitative exploratory and descriptive study will be conducted using individual interviews (clinicians and health care managers) and focus groups (participants).

The successful implementation of this project will bring a unique experience in Quebec of implementing telerehabilitation in a health care facility. The CIUSSS de l'Estrie-CHUS could become a leader in sharing its experience for large-scale implementation in Quebec. The application in orthopedic outpatient clinics may be generalized to other clientele by increasing accessibility to rehabilitation services for clients where accessibility is an issue

ELIGIBILITY:
Inclusion Criteria:

* To present a non-urgent condition (status determined during the initial evaluation at the clinic)
* To be apt to understand simple statement
* To have access to internet at and possess an electronic tablet or a computer at

Exclusion Criteria:

* Do not understand French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Change in pain through time | Day 0, 1 month
  0-10 pain scale (0= no pain, 10 = worst pain)

SECONDARY OUTCOMES:
Change in quality of life through time | Day 0, 12 months
  Evaluate quality of life related to physical and mental state (Questionnaire SF-6Dv2 (Health Utility Survey)). This questionnaire provide a multidimensional generic measure of health-related quality of life. In its current form, this questionnaire includes six questions on different aspects of physical and mental health. The score will be converted to QALY (quality-adjusted life year).The cost-utility analysis (CUA) is an increasingly used method to help health decision-maker. The CUA uses the Quality Adjusted Life Years (QALY) that combines the length of life with the health related quality of life (HRQoL) into a single score.
Direct and indirect costs related to intervention | 12 months
  Indirect and direct costs related to intervention. Direct costs are the costs that are essentials for clinical follow-up and refer to the physiotherapists salary and the acquisition of technological equipment (tablet or computer) used by the patient. Indirect costs are needed to optimize the performance of clinical follow-up and take into account the patient's expenses and / or any other necessary expenses related to his/her participation in the RT program. A home-made questionnaire will be administered to collect information about costs.
Satisfaction with service received | 1 month
  Questionnaire about satisfaction of health care received. The satisfaction construct is determined by three distinct factors which include satisfaction with:
  1) the therapist relationship, 2) the services provided, and 3) the organization of services. This tool includes 26 questions, scored on a four-point Likert scale. The total score is calculated based on average satisfaction for the three factors, with higher scores indicating higher levels of satisfaction (on a 0-100 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Tousignant, Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Research Center on Aging, Sherbrooke, Quebec
  - Research Centre on Aging, Sherbrooke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Renard M, Gaboury I, Michaud F, Tousignant M. The acceptability of two remote monitoring modalities for patients waiting for services in a physiotherapy outpatient clinic. Musculoskeletal Care. 2022 Sep;20(3):616-624. doi: 10.1002/msc.1622. Epub 2022 Feb 10. PMID 35142425